CLINICAL TRIAL: NCT00373451
Title: Randomized, Double-Blind, Active-Controlled, Multicenter Trial of Abciximab And Bivalirudin in Patients With Non-ST-Segment Elevation Myocardial Infarction Undergoing Percutaneous Coronary Interventions (ISAR-REACT-4)
Brief Title: Randomized Comparison of Abciximab Plus Heparin With Bivalirudin in Acute Coronary Syndrome
Acronym: ISAR-REACT-4
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GE IDE No. A01106
Record Dates: First submitted 2006-09-07; First posted 2006-09-08 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: Myocardial Infarction; Coronary Disease
Keywords: NSTEMI
MeSH Terms: conditions — Myocardial Infarction; Coronary Disease; Non-ST Elevated Myocardial Infarction | interventions — Abciximab; bivalirudin; Heparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Abciximab+UFH (Experimental): Abciximab and unfractionated heparin as bolus given during PCI and abciximab-perfusion for 12 hours after PCI
  Interventions: Drug: Abciximab + UFH; Drug: Heparin
- Bivalirudin (Active Comparator): Bivalirudin given only during PCI
  Interventions: Drug: Bivalirudin

INTERVENTIONS:
Drug: Abciximab + UFH — Abciximab (0.25 mg/kg of body weight bolus, followed by a 0.125 µg/kg/minute [maximum of 10 µg/minute] infusion for 12 hours)
  Other Names: ReoPro
  Arms: Abciximab+UFH
Drug: Bivalirudin — Bivalirudin (intravenous bolus of 0.75 mg/kg prior to the start of the intervention, followed by infusion of 1.75 mg/kg per hour for the duration of the procedure)
  Other Names: Angiox
  Arms: Bivalirudin
Drug: Heparin — i.v. bolus of 70 units/kg/body weight of unfractionated heparin
  Other Names: unfractionated heparin
  Arms: Abciximab+UFH

SUMMARY:
The purpose of this study is to determine which of these anti-clotting medications, abciximab plus unfractionated heparin or bivalirudin, is more effective to prevent thrombotic and bleeding complications in patients suffering from a heart attack and undergoing coronary intervention.

DETAILED DESCRIPTION:
Non-ST elevation myocardial infarction (NSTEMI) is associated with an increased risk of death and is a major reason for hospital admissions. Most frequently, the sequence of events that leads to NSTEMI is characterized by a disrupted atherosclerotic plaque, platelet activation and aggregation, thrombus formation and microembolizations. Patients with NSTEMI are treated with an early invasive strategy and there is intensive work in progress to define the optimal antithrombotic therapy to be used in adjunct to percutaneous coronary intervention (PCI) in these patients. Bivalirudin, a direct thrombin inhibitor, and the glycoprotein IIb/IIIa inhibitor (GPI) abciximab have been in the focus of recent trials in patients with acute coronary syndrome (ACS). In a recent randomized, open-label trial (ACUITY trial), patients with the suspicion of ACS on the basis of the type of anginal symptoms, ST-segment displacement, elevated biomarkers or several risk indicators were randomized to receive bivalirudin alone with bail-out GPIs, bivalirudin plus GPIs, or heparin/low-molecular weight heparin plus a GPI. The GPIs most frequently used were eptifibatide and tirofiban. Abciximab was given in only < 9% of the cases. In another randomized, double-blind, placebo-controlled trial (ISAR-REACT-2) including ACS patients undergoing PCI, abciximab was administered in cath lab and was associated with a significant reduction of ischemic events in patients with NSTEMI, and did not lead to a measurable increase in major bleeding complications. However, it is not known whether abciximab is also superior to bivalirudin in patients with NSTEMI. We designed this study to assess whether abciximab added to unfractionated heparin is superior to bivalirudin in patients with NSTEMI.

ELIGIBILITY:
Inclusion Criteria:

* Episode of unstable angina
* Elevated cardiac markers
* Angiographic lesions requiring PCI
* Informed, written consent

Exclusion Criteria:

* Age < 18 years and > 80 years
* ST-segment elevation acute myocardial infarction within 48 hours
* Cardiogenic shock
* Pericarditis
* Malignancies or other comorbid conditions with life expectancy less than one year or that may result in protocol non-compliance
* Active bleeding; bleeding diathesis; history of gastrointestinal or genitourinary bleeding, recent trauma or major surgery in the last month; history of intracranial bleeding or structural abnormalities; suspected aortic dissection; pericarditis; and patient's refusal to blood transfusion
* Oral anticoagulation therapy with coumarin derivative within the last 7 days
* Recent use of GPIIb/IIIa inhibitors within 14 days
* Treatment with unfractionated heparin within 4 hours unless ACT > 150sec; or low-molecular weight heparin within 8 hours before randomization
* Treatment with bivalirudin within 24 hours before randomization
* Severe uncontrolled hypertension > 180/110 mm Hg unresponsive to therapy
* Planned staged PCI procedure within 30 days from index procedure or prior PCI within the last 30 days
* Relevant hematologic deviations
* Glomerular filtration rate (GFR) < 30 ml/min or serum creatinine > 30 mg/L or dependence on renal dialysis
* Known allergy or intolerance to the study medications, stainless steel or true anaphylaxis after prior exposure to contrast media
* Previous enrollment in this trial
* Women who are known to be pregnant, who are of childbearing potential and test positive for pregnancy, who have given birth within the last 90 days, who are breastfeeding
* Patient's inability to fully cooperate with the study protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1721 (Actual)
Dates: Start 2006-07; Primary Completion 2011-05 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Composite of death, large recurrent myocardial infarction (MI), urgent target vessel revascularization (TVR) or major bleeding | 30 days

SECONDARY OUTCOMES:
Composite end point of death, any recurrent myocardial infarction or urgent TVR | 30 days
Major bleedings | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Albert Schoemig, MD, Study Chair — Deutsches Herzzentrum Muenchen; Adnan Kastrati, MD, Principal Investigator — Deutsches Herzzentrum Muenchen
Locations (9):
- Germany (8):
  - Herz-Zentrum Bad Krozingen, Bad Krozingen
  - Herz- und Gefaessklinik, Kardiologie, Bad Neustadt an der Saale
  - Vivantes Klinikum im Friedrichshain, Berlin
  - Vivantes Auguste Viktoria Klinikum, Berlin
  - Vivantes Klinikum Neukoelln, Berlin
  - Deutsches Herzzentrum Muenchen, Munich
  - Medizinische Klinik, Klinikum rechts der Isar, München
  - Marienhospital Osnabrueck, Osnabrück
- Ospedale Cageggi, Florence, Italy

REFERENCES:
- [Background] Braunwald E, Antman EM, Beasley JW, Califf RM, Cheitlin MD, Hochman JS, Jones RH, Kereiakes D, Kupersmith J, Levin TN, Pepine CJ, Schaeffer JW, Smith EE 3rd, Steward DE, Theroux P, Gibbons RJ, Alpert JS, Faxon DP, Fuster V, Gregoratos G, Hiratzka LF, Jacobs AK, Smith SC Jr; American College of Cardiology; American Heart Association. Committee on the Management of Patients With Unstable Angina. ACC/AHA 2002 guideline update for the management of patients with unstable angina and non-ST-segment elevation myocardial infarction--summary article: a report of the American College of Cardiology/American Heart Association task force on practice guidelines (Committee on the Management of Patients With Unstable Angina). J Am Coll Cardiol. 2002 Oct 2;40(7):1366-74. doi: 10.1016/s0735-1097(02)02336-7. No abstract available. PMID 12383588
- [Background] Schulman SP. Antiplatelet therapy in non-ST-segment elevation acute coronary syndromes. JAMA. 2004 Oct 20;292(15):1875-82. doi: 10.1001/jama.292.15.1875. PMID 15494586
- [Background] Neumann FJ, Kastrati A, Pogatsa-Murray G, Mehilli J, Bollwein H, Bestehorn HP, Schmitt C, Seyfarth M, Dirschinger J, Schomig A. Evaluation of prolonged antithrombotic pretreatment ("cooling-off" strategy) before intervention in patients with unstable coronary syndromes: a randomized controlled trial. JAMA. 2003 Sep 24;290(12):1593-9. doi: 10.1001/jama.290.12.1593. PMID 14506118
- [Background] Silber S, Albertsson P, Aviles FF, Camici PG, Colombo A, Hamm C, Jorgensen E, Marco J, Nordrehaug JE, Ruzyllo W, Urban P, Stone GW, Wijns W; Task Force for Percutaneous Coronary Interventions of the European Society of Cardiology. Guidelines for percutaneous coronary interventions. The Task Force for Percutaneous Coronary Interventions of the European Society of Cardiology. Eur Heart J. 2005 Apr;26(8):804-47. doi: 10.1093/eurheartj/ehi138. Epub 2005 Mar 15. PMID 15769784
- [Background] Kastrati A, Mehilli J, Neumann FJ, Dotzer F, ten Berg J, Bollwein H, Graf I, Ibrahim M, Pache J, Seyfarth M, Schuhlen H, Dirschinger J, Berger PB, Schomig A; Intracoronary Stenting and Antithrombotic: Regimen Rapid Early Action for Coronary Treatment 2 (ISAR-REACT 2) Trial Investigators. Abciximab in patients with acute coronary syndromes undergoing percutaneous coronary intervention after clopidogrel pretreatment: the ISAR-REACT 2 randomized trial. JAMA. 2006 Apr 5;295(13):1531-8. doi: 10.1001/jama.295.13.joc60034. Epub 2006 Mar 13. PMID 16533938
- [Derived] Mehilli J, Neumann FJ, Ndrepepa G, King L, Schulz S, Maimer Rodrigues da Cunha F, Jochheim D, Byrne RA, Hausleiter J, Ott I, Massberg S, Kastrati A, Pache J. Sex-related effectiveness of bivalirudin versus abciximab and heparin in non-ST-segment elevation myocardial infarction. Am Heart J. 2013 Apr;165(4):537-43. doi: 10.1016/j.ahj.2012.12.021. Epub 2013 Feb 19. PMID 23537970
- [Derived] Schulz S, Kastrati A, Ferenc M, Massberg S, Birkmeier KA, Laugwitz KL, Kufner S, Gick M, Dommasch M, Schuhlen H, Schomig A, Berger PB, Mehilli J, Neumann FJ; Intracoronary Stenting and Antithrombotic Regimen: Rapid Early Action for Coronary Treatment (ISAR-REACT) 4 Trial Investigators. One-year outcomes with abciximab and unfractionated heparin versus bivalirudin during percutaneous coronary interventions in patients with non-ST-segment elevation myocardial infarction: updated results from the ISAR-REACT 4 trial. EuroIntervention. 2013 Aug 22;9(4):430-6. doi: 10.4244/EIJV9I4A71. PMID 23455033
- [Derived] Ndrepepa G, Neumann FJ, Deliargyris EN, Mehran R, Mehilli J, Ferenc M, Schulz S, Schomig A, Kastrati A, Stone GW. Bivalirudin versus heparin plus a glycoprotein IIb/IIIa inhibitor in patients with non-ST-segment elevation myocardial infarction undergoing percutaneous coronary intervention after clopidogrel pretreatment: pooled analysis from the ACUITY and ISAR-REACT 4 trials. Circ Cardiovasc Interv. 2012 Oct;5(5):705-12. doi: 10.1161/CIRCINTERVENTIONS.112.972869. Epub 2012 Oct 9. PMID 23048052
- [Derived] Sibbing D, Bernlochner I, Schulz S, Massberg S, Schomig A, Mehilli J, Kastrati A. The impact of smoking on the antiplatelet action of clopidogrel in non-ST-elevation myocardial infarction patients: results from the ISAR-REACT 4 platelet substudy. J Thromb Haemost. 2012 Oct;10(10):2199-202. doi: 10.1111/j.1538-7836.2012.04867.x. No abstract available. PMID 22845802
- [Derived] Sibbing D, Bernlochner I, Schulz S, Massberg S, Schomig A, Mehilli J, Kastrati A. Prognostic value of a high on-clopidogrel treatment platelet reactivity in bivalirudin versus abciximab treated non-ST-segment elevation myocardial infarction patients. ISAR-REACT 4 (Intracoronary Stenting and Antithrombotic Regimen: Rapid Early Action for Coronary Treatment-4) platelet substudy. J Am Coll Cardiol. 2012 Jul 31;60(5):369-77. doi: 10.1016/j.jacc.2012.02.044. Epub 2012 Jun 6. PMID 22682553
- [Derived] Kastrati A, Neumann FJ, Schulz S, Massberg S, Byrne RA, Ferenc M, Laugwitz KL, Pache J, Ott I, Hausleiter J, Seyfarth M, Gick M, Antoniucci D, Schomig A, Berger PB, Mehilli J; ISAR-REACT 4 Trial Investigators. Abciximab and heparin versus bivalirudin for non-ST-elevation myocardial infarction. N Engl J Med. 2011 Nov 24;365(21):1980-9. doi: 10.1056/NEJMoa1109596. Epub 2011 Nov 13. PMID 22077909